CLINICAL TRIAL: NCT03302286
Title: Effects of Extra Corporeal Circuit Prime on Electrolytes Balance and Clinical Outcome Following Cardiac Surgery
Acronym: Prime
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Region Skane (Other)
Responsible Party: Principal Investigator, Snejana Hyllén, MD, Region Skane
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: 2017/422
Record Dates: First submitted 2017-09-25; First posted 2017-10-05 (Actual); Last update posted 2022-01-18 (Actual); Status verified 2022-01

CONDITIONS: Cardiac Surgery
Keywords: Heart-Lung Machine; Cardiopulmonary Bypass

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mannitol Prime (Active Comparator): This group will undergo cardiac surgery with heart-lung machine with priming solution of Ringer's acetate 1000 ml, Mannitol 200 ml, Heparin 10000 units and 80 mmol sodium.
  Interventions: Diagnostic Test: Heart-lung machine primining solution which includes Mannitol
- NonMannitol Prime (Active Comparator): This group will receive a priming solution of Ringer´s acetate 1200 ml, Heparin 10000 units and 80 mmol sodium.
  Interventions: Diagnostic Test: Heart-lung machine primining solution which does not include Mannitol

INTERVENTIONS:
Diagnostic Test: Heart-lung machine primining solution which includes Mannitol — This study group will undergo cardiopulmonary bypass with priming solution of Ringer's acetate 1000 ml, Mannitol 200 ml, Heparin 10000 units and 80 mmol sodium.
  Arms: Mannitol Prime
Diagnostic Test: Heart-lung machine primining solution which does not include Mannitol — This study group will undergo cardiopulmonary bypass with priming solution of Ringer's acetate 1200 ml, Heparin 10000 units and 80 mmol sodium.
  Arms: NonMannitol Prime

SUMMARY:
About 6000 heart operations are performed in Sweden every year. A heart-lung machine is used almost exclusively in all heart operations. This machine fills the role of heart and lungs during surgery while the heart is stopped. The extra corporeal circuit (ECC) prime results in hemodilution, as assessed from the decrease in haematocrit, electrolyte concentration and total protein content. This hemodilution is an unavoidable consequence of the use of a heart-lung machine with nonblood ECC prime. The alteration of the patient´s blood volume and electrolytes is affected by the prime solution and can be maintained within normal limits. There are no clear recommendation regarding prime components and numerous prime solutions are in use worldwide.

The aim of this study is to investigate whether the use of mannitol in heart-lung machine prime has an effect on electrolytes levels and osmolality when compared with patients who receive no Mannitol.

ELIGIBILITY:
Inclusion Criteria:

* adult patients of both sexes who will undergo elective isolated coronary artery bypass grafting at the Department of Cardiothoracic Surgery, Skåne University Hospital, Lund

Exclusion Criteria:

* heart failure with left ventricular ejection fraction below 50%
* small size (defined as bodyweight less than 50 kg)
* anaemia with haematocrit less than 24%
* patients with previous cardiac surgery
* patients who receive other fluids or more than 1000 ml additional Ringers's Acetate during cardiopulmonary bypass
* patients with peroperative complications including massive peroperative fluid transfusions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2017-10-01 (Actual); Primary Completion 2021-10-01 (Actual); Study Completion 2021-10-01 (Actual)

PRIMARY OUTCOMES:
osmolality | Measurements will be taken three minutes after administration of cardioplegia during cardiopulmonary bapass.
  This study uses blood samples that are taken at predefined timepoints.

SECONDARY OUTCOMES:
urine outcome | Measurements will be taken during first 24 hours following cardiac surgery
  Production of urine will be studed following cardiac operation

CONTACTS AND LOCATIONS:
Overall Officials: Snejana Hyllen, phd, Principal Investigator — Region Skane
Locations (1):
- Thorax, Lund, Skåne County, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Skold A, Dardashti A, Lindstedt S, Hyllen S. No benefit of adding mannitol to cardiopulmonary bypass priming solution assessing cystatin C. A randomized clinical trial. Perfusion. 2025 May 24:2676591251344857. doi: 10.1177/02676591251344857. Online ahead of print. PMID 40411794